CLINICAL TRIAL: NCT00277862
Title: Role of Rapid Virologic Response in Determining Treatment Duration of Peginterferon Alfa-2b/Ribavirin in Chronic Hepatitis C Genotype 4
Brief Title: Pegylated Interferon and Ribavirin Therapy in Chronic Hepatitis Genotype 4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Schering-Plough (Industry); Fulbright (Other); Tempus AI (Industry); International Society for Infectious Diseases (Other)
Responsible Party: Dr. Nelly Sedky, Dr. Gehan Galal, DIAGSERA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G43230832638
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-02

CONDITIONS: Hepatitis C
Keywords: chronic hepatitis C;; peg-interferon alfa-2b;; ribavirin,; rapid virologic response,; sustained virological response
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): 1. Pegylated IFN- alpha 2b
  2. Ribavirin for 24 weeks (patients with RVR)
  Interventions: Drug: Pegylated IFN- alpha 2b; Drug: Ribavirin
- 2 (Active Comparator): 1. Pegylated IFN- alpha 2b
  2. Ribavirin for 36 weeks (patients with complete EVR)
  Interventions: Drug: Pegylated IFN- alpha 2b; Drug: Ribavirin
- 3 (Active Comparator): 1. Pegylated IFN- alpha 2b
  2. Ribavirin for 48 weeks (patients with partial EVR)
  Interventions: Drug: Pegylated IFN- alpha 2b; Drug: Ribavirin
- 4 (Active Comparator): 1. Pegylated IFN- alpha 2b
  2. Ribavirin for 48 weeks (control)
  Interventions: Drug: Pegylated IFN- alpha 2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated IFN- alpha 2b
  Other Names: PEG-IFN alpha-2b; PEG-Intron™
Drug: Ribavirin
  Other Names: Rebetol; Virin; Ribavrin

SUMMARY:
Genotype 4 is the least-studied hepatitis C virus genotype and was considered a difficult to treat genotype due to the disappointing response of chronic hepatitis C genotype 4 to conventional interferon monotherapy. Recent reports showed that pegylated interferon and ribavirin combination therapy markedly increased the SVR rate to 55-70%. The duration of treatment has not been accurately defined. The main objective of this is to assess the duration of pegylated interferon ribavirin therapy in chronic hepatitis genotype 4 and assess the clinical utility of rapid and early virologic response in determining the optimal duration of peg interferon ribavirin therapy in chronic hepatitis C.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) genotype 4 is the most frequent cause of chronic hepatitis C in Middle East, North Africa and sub-Saharan Africa. In countries like Egypt, 73 to 90% of cases of chronic hepatitis C are caused by genotype 4. Recently, epidemiological reports showed spread of HCV-4 infection in Western countries such as France, Italy, Greece, Spain and the United States particularly among intravenous drug users.

Genotype 4 is the least-studied hepatitis C virus genotype and was considered a difficult to treat genotype due to the disappointing response of chronic hepatitis C genotype 4 to conventional interferon monotherapy. Recent reports showed that pegylated interferon and ribavirin combination therapy markedly increased the SVR rate to 55-70%. We have previously shown that, treatment patients with chronic HVCG4with PEG-IFN α-2b plus ribavirin for 36 or 48 weeks was more effective (SVR 66% and 69%, respectively) than for 24 weeks.

It has been shown in previous studies on chronic hepatitis C genotype 1 that individuals who achieve an early virologic have a higher chance to achieve a sustained virologic response. Peg interferon and ribavirin therapy is associated with adverse events and is expensive; therefore, careful determination of the optimal treatment duration is crucial as it spares the patient unnecessary or prolonged therapy and enhances the cost-effectiveness of therapy.

Therefore the main objective of this randomized, multicenter trial is to assess the clinical utility of rapid and early virologic response in determining the optimal duration of peg interferon ribavirin therapy in chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:Adult males and females, 18 to 50 years of age; with documented chronic hepatitis C according to the following criteria: elevated serum alanine aminotransferase (ALT) above the upper limit of normal (40 U/l) on two occasions during the preceding six months; anti-HCV positive anti-body status assessed by second generation enzyme linked immunosorbent assay (Roche Diagnostics, Branchburg, New Jersey, USA); positive polymerase chain reaction for HCV RNA (Cobas Amplicor HCV Monitor v2.0; lower limit of quantitation 50 IU/mL); genotype 4; and criteria for chronic hepatitis C in liver biopsy performed within the preceding year with no signs of cirrhosis or bridging fibrosis on pretreatment liver biopsy.

-

Exclusion Criteria:

* Previous IFN-alpha therapy; other liver diseases such as hepatitis A, hepatitis B, schistosomiasis, autoimmune hepatitis, alcoholic liver disease, drug induced hepatitis, or decompensated liver disease; coinfection with schistosomiasis or human immunodeficiency virus; neutro¬penia (,1 500/mm3); thrombocytopenia (,90 000/mm3); creatinine concentration .1.5 times the upper limit of normal; serum a fetoprotein concentration .25 ng/ml; organ transplant; neoplastic disease; severe cardiac or pulmonary disease; unstable thyroid dysfunction; psychiatric disorder; current pregnancy or breast feeding; or therapy with immunomodulatory agents within the last six months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2002-04; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
sustained virologic response defined as undetectable serum HCV RNA levels (Amplicor HCV, Roche Molecular Systems; lower limit of detection (LLD) of 50 IU/mL) | 18 months

SECONDARY OUTCOMES:
Virologic response at the end of treatment (EOT) defined as undetectable HCV RNA serum levels (50 IU/ml) at the end of the scheduled treatment period | 6-12 months and 6 months follow-up
sustained virologic response (primary) histological response (secondary) biochemical response (secondary) | 6-12 months treatment), 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sanaa M Kamal, M.D.; Ph.D, Principal Investigator — AUS Specialized Hospital, Cairo, Cairo, 11351, Egypt;; Amany Sayed Ahmad, M.D., Principal Investigator — DIAGSERA; Samer El Kamary, Principal Investigator — UMB; Amal Abdel Baky, M.D., Principal Investigator — DIGSERA
Locations (4):
- Egypt (4):
  - AUS Specialized Hospital,, Cairo, Cairo Governorate
  - DIACSERA, Cairo
  - MISR Welding, Cairo
  - ELectricity Auth, Mynia and Cairo

REFERENCES:
- [Background] Kamal SM, El Tawil AA, Nakano T, He Q, Rasenack J, Hakam SA, Saleh WA, Ismail A, Aziz AA, Madwar MA. Peginterferon alpha-2b and ribavirin therapy in chronic hepatitis C genotype 4: impact of treatment duration and viral kinetics on sustained virological response. Gut. 2005 Jun;54(6):858-66. doi: 10.1136/gut.2004.057182. PMID 15888797
- [Background] Kamal SM, Fehr J, Roesler B, Peters T, Rasenack JW. Peginterferon alone or with ribavirin enhances HCV-specific CD4 T-helper 1 responses in patients with chronic hepatitis C. Gastroenterology. 2002 Oct;123(4):1070-83. doi: 10.1053/gast.2002.36045. PMID 12360469
- [Derived] Kamal SM, El Kamary SS, Shardell MD, Hashem M, Ahmed IN, Muhammadi M, Sayed K, Moustafa A, Hakem SA, Ibrahiem A, Moniem M, Mansour H, Abdelaziz M. Pegylated interferon alpha-2b plus ribavirin in patients with genotype 4 chronic hepatitis C: The role of rapid and early virologic response. Hepatology. 2007 Dec;46(6):1732-40. doi: 10.1002/hep.21917. PMID 17943989